CLINICAL TRIAL: NCT04235972
Title: Evaluation of Staple Watson Wrist Arthrodesis
Acronym: ESWWA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 35RC19_8861; 2019-A01553-54 (Other: Id-RCB)
Record Dates: First submitted 2019-12-26; First posted 2020-01-22 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Osteoarthritis Wrist
Keywords: orthopaedic surgery; Staples

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arthrodesis surgery patients (Other): A follow-up consultation is organized which includes: A clinical examination with standard data collection as well as a face and profile radiograph of the operated wrist.
  Interventions: Other: Follow-up consultation

INTERVENTIONS:
Other: Follow-up consultation — A follow-up consultation is organized which includes: A clinical examination with standard data collection as well as a face and profile radiograph of the operated wrist.

SUMMARY:
When the wrist is damaged, for traumatic or degenerative reasons, the cartilage is worn out and the bones rub together: this is osteoarthritis. In order to stop this pain, it may be necessary to block these bones from each other, sacrificing mobility to achieve indolence.

Multiple techniques are described according to the type of osteoarthritis and for each type of osteoarthritis itself, but the principle remains the same. The methods currently commonly proposed are the staple and the screwed plate.

The aim of the study is to evaluate the surgical practice of the Orthopaedics and Traumatology department of the University Hospital of Rennes, and its long-term results, as this type of surgery is intended to be definitive.

DETAILED DESCRIPTION:
The surgery performed in the Orthopaedics and Traumatology department of the University Hospital of Rennes, has 2 notable points: its technique and its equipment.

* The procedure is based on the staples 4Fusion1 (Stryker/Memometal), which is still poorly assessed in the literature.
* The surgical procedure has several technical specificities: intra osseous cartilage freshening and preservation of the lunotriquetral ligament if intact.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients
* All patients operated on for a 4-bones arthrodesis performed by stapling at the CHU RENNES between 1 January 2008 and 31 December 2017 with 4fusion stapling
* Patients who gave consent after full information

Exclusion Criteria:

* Refusal to participate after information
* Protected adults
* Person deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-01-07 (Actual)

PRIMARY OUTCOMES:
Assessment of the surgical procedure | Day 1
  Assessement of the bones consolidation at at least 6 weeks post-surgery, using a radiological criterion : 3 out of 4 line spacing merged

SECONDARY OUTCOMES:
Pain assessment | Day 1
  Evolution in pain reported by the patient by a pain assessment scale, with reference to preoperative assessment.
  Evaluation is based on the visual analog scale (VAS) in which the patients select a whole number (0-10 integers) that best reflects the intensity of their pain
Grip force | Day 1
  Change of the grip force measured by Jamar's hydraulic dynamometer, compared to pre-operative assessment
Functional assessment of the wrist with Mayo Wrist Score | Day 1
  International validated functional score. This evaluation yields a total score out of 100 points qualified as poor if <65 up to Excellent if >90.
Functional assessment of the wrist with Quick Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire | Day 1
  International validated functional score. The Quick DASH tool uses a 5-point Likert scale from which the patient can select an appropriate number corresponding to his/her severity level/ function level
Functional assessment of the wrist with Patient-Rated Wrist Evaluation | Day 1
  International validated functional score. The Patient-Rated Wrist Evaluation (PRWE) allows patients to rate their levels of wrist pain and disability from 0 to 10
Patient's overall satisfaction about surgery | Day 1
  Patient's overall satisfaction assessed by the question: "Would you do the surgery again? (balance between 0 and 10)"
Material hindrance | Day 1
  Specific items assessed during clinical evaluations. Quoted as 1 if at least one of the following events is evoked : Material-related pain, skin irritation, re-intervention for remote ablation
Mean mobility arc | Day 1
  Measurement of the arc of mobility in flexion - extension by goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Warren KIM, MD, Study Director — CHU Rennes
Locations (1):
- CHU de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mevel G, De Geyer A, Kim W, Ebalard M, Ropars M, Dreano T. Four-corner arthrodesis using the 4Fusion(R) quadripodal shape memory staple: a long-term review. J Hand Surg Eur Vol. 2022 Apr;47(4):387-392. doi: 10.1177/17531934211063614. Epub 2021 Dec 1. PMID 34851782